CLINICAL TRIAL: NCT06651320
Title: Effect of Preoperative Patient Education Via Animated Videos in Patients Undergoing Operative Hysteroscopy Under Anesthesia
Brief Title: Preoperative Animated Videos in Patients Undergoing Operative Hysteroscopy Under Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Matan Mor, Attending physician - Minimal Invasive Gynecology Unit, Shamir Medical Center, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ASF-189-24
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Satisfaction with Care
Keywords: hysteroscopy
MeSH Terms: conditions — Anxiety Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 Intervention group: traditional patient education (nurse + physician pre-procedural counseling) + (Experimental): intervention
  Interventions: Other: The patients in the interventional arm will be introduced to video will be introduced to a concise, animated video explaining the steps they are about to undergo in the department, the OR, recovery
- 2 The Nonintervention group would receive the traditional patient education before the procedure (vi (No Intervention)

INTERVENTIONS:
Other: The patients in the interventional arm will be introduced to video will be introduced to a concise, animated video explaining the steps they are about to undergo in the department, the OR, recovery — The patients in the interventional arm will be introduced to video will be introduced to a concise, animated video explaining the steps they are about to undergo in the department, the OR, recovery and discharge. How to prepare for the procedure, what to expect during and after the procedure and what are the possible follow up scenarios.
  In order to overcome language berries videos would be available in basic 6th grader language and translated into English, Arabic and Russian for the non-Hebrew speaking population.
  There would be one staff member aware of the patient's allocation the international Vs nonintervention arm while the rest of the staff would be masked to the research arm the patient was allocated to.
  Once they have watched the video they would be asked to fill up a questionnaire their anxiety level concerning the procedure (STAI-S).
  Arms: 1 Intervention group: traditional patient education (nurse + physician pre-procedural counseling) +

SUMMARY:
The goal of this clinical trial is to assess if the use of an audiovisual animated video, describing the gynecological procedure (hysteroscopy) the patient is about to undergo, will help to reduce the patient's level of anxiety, affect her anesthesia parameters and increase their overall satisfaction from the procedure.

Our hypothesis is that patient who will watch the video (intervention group) will experience less anxiety, will have lower heart rate and lower blood pressure during the procedure, and have overall more satisfaction with the procedure, compared to patients who will not watch the preoperative video (control group).

Patients will be asked to rate their anxiety level before the procedure and their satisfaction afterwards.

DETAILED DESCRIPTION:
Is has been questioned what the effectiveness of various modes of delivering preoperative education in reducing preoperative anxiety is and as a result pain and overall satisfaction of patients from surgical producers. It is known that women undergoing hysteroscopy suffer from significant levels of anxiety, with repercussions on pain perception, success rates and satisfaction (1). In the inpatient surgery setting, preoperative anxiety is commonly managed by means of pharmacological interventions such as the use of anxiolytics and sedatives. Communication and patient education have been proved as effective tools to reduce preoperative anxiety, and their role should be increasingly acknowledged, now that many patients are active consumers of unfiltered and largely unreliable information through the Internet.

One meta-analysis which included 14 interventional trials (1) concluded that preoperative education interventions are promising in reducing preoperative anxiety in patients scheduled for surgical procedures (1).

Objective To assess if the use of an audiovisual animated video describing the gynecological procedure (hysteroscopy) the patient is about to undergo will help to reduce the patient's level of anxiety, affect her anesthesia parameters and increase their overall satisfaction from the procedure.

Design A randomized control trial including the patients undergoing operative hysteroscopy under anesthesia in the operation room via the endoscopy unit's team, Shamir hospital, Israel.

Inclusion criteria: adult patients (above 18 and older), undergoing operative hysteroscopy under anesthesia in our OR due to uterine findings previously diagnosed during diagnostic hysteroscopy.

Exclusion criteria: Patients who patient who are not able to watch the audiovisual video or who cannot sign a consent form.

The research would require a total 100 patients. The sample sign is based upon a previous study done in our institute assessing the effect of an audiovisual video on anxiety levels of patients undergoing diagnostic and operative hysteroscopy without anesthesia.

The patients would be randomly divided into the Intervention and Nonintervention group. Patients would be requested to fill up a questionnaire

1. Intervention group: traditional patient education (nurse + physician pre-procedural counseling) + supplemental animation video describing the procedure itself and what to expect from it. This group will receive a code they ca scan so they can watch the video before entering the examination room where the physician will see them and where the hysteroscopy will be performed.
2. The Nonintervention group would receive the traditional patient education before the procedure (via the team's nurse and the doctor performing the procedure) and would be unaware of the animation video in order to avoid bias in the questionnaire.

The patients in the interventional arm will be introduced to video will be introduced to a concise, animated video explaining the steps they are about to undergo in the department, the OR, recovery and discharge. How to prepare for the procedure, what to expect during and after the procedure and what are the possible follow up scenarios.

In order to overcome language berries videos would be available in basic 6th grader language and translated into English, Arabic and Russian for the non-Hebrew speaking population.

There would be one staff member aware of the patient's allocation the international Vs nonintervention arm while the rest of the staff would be masked to the research arm the patient was allocated to.

Once they have watched the video they would be asked to fill up a questionnaire their anxiety level concerning the procedure (STAI-S).

For each patient the performing physician would fill up a basic demographic questionnaire (age, weight, obstetrical history, chronic diseases and medications) and after completing the procedure - information regarding the intrauterine findings and the procedure itself (actual finding, size and location of the finding, procedural length, instruments used, etc).

Anesthesia parameters during the operative hysteroscopy would also be measured including the patients' blood pressure, pulse and BIS and amount of anesthetic agents in order to assess the anesthesia.

In the context of anesthesia, PSI (Patient state Index) is a monitoring tool used to assess the depth of anesthesia in patients during surgery. It helps anesthesiologists ensure that a patient is neither too deeply nor too lightly anesthetized, aiming for an optimal balance. It uses sensors placed on the patient's forehead to measure electrical activity in the brain (EEG) and processes these signals and calculates a PSI value between 0-100. Score of 25-50 is the target range for general anesthesia, suggesting an adequate depth of anesthesia where the patient is unlikely to be conscious or aware. 50< may indicate a lighter plane of anesthesia where there is a risk of consciousness while 100 means fully awake and alert. By monitoring BIS, anesthesiologists can adjust the amount of anesthetic agents in real-time to maintain appropriate anesthesia levels, avoiding both under-dosing (which can lead to awareness) and over-dosing (which can cause prolonged recovery times or side effects). PSI is used alongside other clinical assessments and monitoring devices, such as heart rate and blood pressure, to guide anesthesia management.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (above 18 and older),
* Patients undergoing operative hysteroscopy under anesthesia in our OR due to uterine findings previously diagnosed during diagnostic hysteroscopy.

Exclusion Criteria:

* Patients who are not able to watch the audiovisual video
* Patients who cannot sign a consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients who experienced anxiety before the procedure as assessed by STAI-S | From the enrollment to the beginning of general anesthesia, up to 48 hours

SECONDARY OUTCOMES:
Heart rate (bpm) | During the procedure, up to 120 minutes
Blood pressure (mmHg) | During the procedure, up to 120 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Shamir Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ayyadhah Alanazi A. Reducing anxiety in preoperative patients: a systematic review. Br J Nurs. 2014 Apr 10-23;23(7):387-93. doi: 10.12968/bjon.2014.23.7.387. PMID 24732993
- [Background] Gambadauro P, Navaratnarajah R, Carli V. Anxiety at outpatient hysteroscopy. Gynecol Surg. 2015;12(3):189-196. doi: 10.1007/s10397-015-0895-3. Epub 2015 May 13. PMID 26283891